CLINICAL TRIAL: NCT00399438
Title: A Dose-Ranging Study of the Pharmacodynamic Effects of BMS-562086 on Gastrointestinal Transit in Women With Diarrhea-Predominant Irritable Bowel Syndrome
Brief Title: A Study of BMS-562086 in Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CN148-013
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: Irritable Bowel Syndrome
Keywords: Diarrhea-predominant irritable bowel syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — pexacerfont

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Other): 0 mg
  Interventions: Drug: Placebo
- 2 (Other): 25 mg
  Interventions: Drug: BMS-562086
- 3 (Other): 100 mg
  Interventions: Drug: BMS-562086

INTERVENTIONS:
Drug: Placebo — Tablets, Oral, once daily, 2 weeks
  Arms: 1
Drug: BMS-562086 — Tablets, Oral, once daily, 2 weeks
  Arms: 2; 3

SUMMARY:
The primary purpose of this study is to evaluate the effects of BMS-562086 on small bowel and colonic transits in female subjects with diarrhea-predominant irritable bowel syndrome (D-IBS)

ELIGIBILITY:
Inclusion Criteria:

* Female subjects with D-IBS symptoms based on Rome II criteria and the subject's responses to the Bowel Disease Questionnaire

Exclusion Criteria:

* Clinically significant prolonged diarrhea with dehydration requiring IV fluid within 60 days prior to baseline visit

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2006-12; Primary Completion 2007-10 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Radioscintigraphy will be used to determine the effects of BMS-562086 on gastrointestinal transit | taken at baseline on nominal study days 3,4, and 5 and post dose on nominal study days 14,15, 16

SECONDARY OUTCOMES:
Daily diary will be used to record the effects of BMS-562086 on bowel patterns and visceral symptoms. | throughout the study
Safety | Safety labs at screening, nominal study days -3, 8, 15, 42, and 70 (discharge). ECGs will be taken at screening, nominal days 5 or 6, 14, and discharge. Vital signs will be taken at screening, on nominal days 3, 4, 5, 7, 8, 10, 11, 42 and discharge
Blood pharmacokinetics | PK samples will be taken on nominal days 8, 14 (serial: predose 0.5, 1, 2, 4, 6, 9 hours post dose), 15 (pre dose and 9 hours post dose), 16, 42 and discharge

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States